CLINICAL TRIAL: NCT03298672
Title: A Randomized, Placebo-Controlled, Double-Blinded, First-in-Human Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (Part A) and Multiple Ascending Doses (Part B) of NDX-1017 in Healthy Young and Elderly Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics Study of NDX-1017
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athira Pharma (Industry)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Biotrial Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NDX-1017-0101-01
Record Dates: First submitted 2017-09-21; First posted 2017-10-02 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Cognition; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NDX-1017 (Experimental): NDX-1017 will be administered via subcutaneous injection
  Interventions: Drug: NDX-1017
- Placebo (Placebo Comparator): Placebo will be administered via subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NDX-1017 — Solution of NDX-1017 for subcutaneous injection
  Arms: NDX-1017
Drug: Placebo — Placebo solution for subcutaneous injection
  Arms: Placebo

SUMMARY:
This Phase 1 randomized, placebo-controlled, double-blinded, first-in-human study will evaluate safety, tolerability, and pharmacokinetics of single and multiple ascending doses of NDX-1017 in healthy young and elderly subjects, and elderly subjects with amnestic mild cognitive impairment (MCI), Alzheimer's disease (mild, mild-to-moderate, or moderate), or mixed dementia with Alzheimer's and vascular components (mild, mild-to-moderate, or moderate).

DETAILED DESCRIPTION:
NDX-1017 is being developed for the treatment of Alzheimer's disease (AD).

This Phase 1 randomized, placebo-controlled, double-blinded, first-in-human study will evaluate safety, tolerability, and pharmacokinetics of single and multiple ascending doses of NDX-1017 in healthy young and elderly subjects, and elderly subjects with mild AD. The study contains the following two parts:

Part A:

A single-ascending dose (SAD) study conducted in an inpatient setting for 3 days in healthy young male and healthy elderly male and female volunteers evaluated in up to 7 dose cohorts to identify the maximum tolerated dose (MTD) within the single dose range studied. Up to 56 subjects (aged 18 to 45 years for young and 60 to 85 years for elderly) may be enrolled in Part A.

Part B:

A multiple ascending dose (MAD) study conducted in an inpatient setting for 10 days in male or female healthy elderly volunteers (aged 60 to 85 years) or subjects with amnestic mild cognitive impairment (MCI), Alzheimer's disease (mild, mild-to-moderate, or moderate), or mixed dementia with Alzheimer's and vascular components (mild, mild-to-moderate, or moderate) (aged 40 to 85 years) in up to 6 dose cohorts that were proven tolerable in the SAD part of the study to identify the MTD within the multiple dose range studied. Up to 44 subjects (aged 40 to 85 years) may be enrolled in Part B.

Subjects will be screened for eligibility within 28 days (or 90 days for amnestic MCI, Alzheimer's Disease, or mixed dementia with Alzheimer's and vascular components) prior to enrollment. Those eligible will be admitted to an inpatient facility for investigational product administration, safety monitoring, and collection of blood or urine for pharmacokinetic evaluations.

ELIGIBILITY:
INCLUSION CRITERIA:

* Generally in good health
* Body mass index (BMI) of ≥ 18.0 and ≤ 30.0 kg/m2 at Screening, with minimum weight of 60 kg. (No BMI upper limit for mild AD and amnestic MCI subjects)
* Male subjects and their partners must be willing to comply with the contraceptive requirements of the study. Only female subjects of non-childbearing potential are eligible for participation.
* [Young subjects] Male subjects must be aged 18 to 45 years (inclusive) at the time of Screening.
* [Healthy elder subjects only] Male and female subjects must be aged 60 to 85 years at the time of screening
* [Amnestic MCI and Alzheimer's Subjects] 9. Patients with Alzheimer's disease, with confirmed diagnosis of amnestic mild cognitive impairment, Alzheimer's disease (mild, mild-to-moderate, or moderate), or mixed dementia with Alzheimer's and vascular components (mild, mild-to-moderate, or moderate).

  1. Either newly diagnosed treatment naïve patients, OR,
  2. Patients who are currently on standard Alzheimer's Disease treatment may be considered for participation if they are not tolerating treatment and/or they are willing and clinically able to tolerate a discontinuation, 14 days for dose titration + 5x half-lives for washout, or 4 weeks (whichever is longer) prior to randomization. For these patients, the screening window will be allowed for up to 90 days prior to randomization to evaluate discontinuation of symptomatic treatment for Alzheimer's disease.

EXCLUSION CRITERIA:

* Any medical condition that requires chronic medication use.
* History of drug and/or alcohol abuse within 12 months prior to Screening.
* History of having taken another investigational drug within 30 days prior to Admission (Day -1).
* Donation of blood or plasma within 30 days prior to dosing.
* Major surgery within 90 days prior to Admission (Day -1) or anticipated surgery during the study.
* Smokers
* [Healthy elderly subjects] Reported changes in cognition and reported history of declines in everyday life in the last year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. | Up to 20 days
  Safety and tolerability of single or multiple ascending doses of NDX-1017 as measured by vital signs and clinical laboratory measurements.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax). | Samples collected at predetermined timepoints within 48 hours post-dose.
  Cmax will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Time to maximum observed plasma concentration (Tmax). | Samples collected at predetermined timepoints within 48 hours post-dose.
  Tmax will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Plasma concentration at the end of the dosing interval (Ctrough). | Samples collected at predetermined timepoints within 48 hours post-dose.
  Ctrough will be determined from the last plasma sample prior to the following dose (MAD only).
Area under the plasma concentration time curve (AUC). | Samples collected at predetermined timepoints within 48 hours post-dose.
  AUC will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Half-life (t1/2). | Samples collected at predetermined timepoints within 48 hours post-dose.
  t1/2 will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Hua, PhD, Study Director — Athira Pharma, Inc.
Locations (1):
- Biotrial Inc., Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hua X, Church K, Walker W, L'Hostis P, Viardot G, Danjou P, Hendrix S, Moebius HJ. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Positive Modulator of HGF/MET, Fosgonimeton, in Healthy Volunteers and Subjects with Alzheimer's Disease: Randomized, Placebo-Controlled, Double-Blind, Phase I Clinical Trial. J Alzheimers Dis. 2022;86(3):1399-1413. doi: 10.3233/JAD-215511. PMID 35180125